CLINICAL TRIAL: NCT00416507
Title: Non Resectable But Non Metastatic Adenocarcinoma of the Exocrine Pancreas Non Resecables. Randomised Phase III: Initial Radiochimiotherapy (5-FU, Cisplatine, 60 GY Radiotherapy) Followed by Gemcitabine Versus Gemcitabine Alone
Brief Title: Gemcitabine With or Without Combination Chemotherapy and Radiation Therapy in Treating Patients With Nonmetastatic Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000453847; FFCD-2000-01; EU-20542; FFCD-SFRO-2000-01
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; SPI-77, liposomal

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: liposomal cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, fluorouracil, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving more than one drug (combination chemotherapy) together with radiation therapy may kill more tumor cells. It is not yet known which treatment regimen is more effective for pancreatic cancer.

PURPOSE: This randomized phase III trial is studying gemcitabine, fluorouracil, cisplatin, and radiation therapy to see how well they work compared to gemcitabine alone in treating patients with nonmetastatic pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with nonresectable, nonmetastatic adenocarcinoma of the pancreas treated with gemcitabine hydrochloride with vs without fluorouracil, cisplatin, and radiotherapy followed by gemcitabine hydrochloride.

Secondary

* Compare the toxicities of these regimens in these patients.
* Compare the objective response (complete, partial, or stable) in patients treated with these regimens.
* Compare the clinical benefit, in terms of general condition and weight maintenance in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to WHO performance status (0 or 1 vs 2), initial treatment (laparotomy with or without bilio-digestive diversion) (yes vs no), and peritoneal cytology (positive vs negative). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV over 15 minutes on days 1-5 and 29-33 and fluorouracil IV continuously on days 1-40. Patients also undergo radiotherapy daily, 5 days a week, for 6 weeks.
* Arm II: Patients receive gemcitabine hydrochloride IV over 15 minutes on day 1. Treatment repeats every 7 days for 7 weeks.

Beginning in week 11 of arm I or week 9 of arm II, patients receive gemcitabine hydrochloride IV over 15 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 190 patients will be accrued for this trial.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* No neuroendocrine or other histologies
* No extra-abdominal metastases
* No hepatic or peritoneal metastases by celioscopy

  * Peritoneal carcinomatous (cytology positive by peritoneal lavage) may be allowed
* Nonresectable disease meeting ≥ 1 of the following criteria:

  * Arterial invasion
  * Mesenteric-portal vein invasion > 15 mm and or less than hemicircumference
  * Satellite adenopathies encompassed in the radiation field

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Bilirubin < 1.75 mg/dL
* Creatinine < 1.5 mg/dL
* WBC > 1,500/mm³
* Platelet count > 100,000/mm³
* No major organ disorder, including cardiac or coronary insufficiency
* Prothrombin time > 80%
* No psychiatric or social condition that would preclude study therapy
* No other malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No contraindications to radiotherapy or chemotherapy
* No intractable pancreatic pain not relieved by morphine and/or analgesic radiotherapy

PRIOR CONCURRENT THERAPY:

* No prior adjuvant or palliative chemotherapy or radiotherapy
* Prior surgical diversion of the biliary and/or digestive tract allowed

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2000-03; Primary Completion 2005-07 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Mornex, MD, PhD, Study Chair — Centre Hospitalier Lyon Sud

REFERENCES:
- [Result] Chauffert B, Mornex F, Bonnetain F, Rougier P, Mariette C, Bouche O, Bosset JF, Aparicio T, Mineur L, Azzedine A, Hammel P, Butel J, Stremsdoerfer N, Maingon P, Bedenne L. Phase III trial comparing intensive induction chemoradiotherapy (60 Gy, infusional 5-FU and intermittent cisplatin) followed by maintenance gemcitabine with gemcitabine alone for locally advanced unresectable pancreatic cancer. Definitive results of the 2000-01 FFCD/SFRO study. Ann Oncol. 2008 Sep;19(9):1592-9. doi: 10.1093/annonc/mdn281. Epub 2008 May 7. PMID 18467316
- [Result] Mornex F, Chauffert B, Bonnetain F, et al.: Definitive results of the French FFCD-SFRO 2000-01 study: phase III trial comparing chemoradiotherapy (cisplatin and infusional 5-FU) followed by gemcitabine vs. gemcitabine alone in patients with locally advanced non metastatic pancreatic cancer. [Abstract] Int J Radiat Oncol Biol Phys 69 (3): A-135, S77, 2007.